CLINICAL TRIAL: NCT06316804
Title: Design and Feasibility of a Mobile Mental Health Stigma Reduction Intervention Among Black Adults With Depression and Anxiety
Brief Title: Mobile Mental Health Stigma Reduction Intervention Among Black Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Aderonke Bamgbose Pederson, Physician, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2022P000580; 1K23MH128535-01A1 (NIH)
Record Dates: First submitted 2024-02-28; First posted 2024-03-18 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Anxiety; Depression; Health Knowledge, Attitudes, Practice; Stigmatization; Mobile Phone Use
Keywords: Stigma; Digital Mental Health; Community Engaged Research; Black Adult; Mobile Health
MeSH Terms: conditions — Anxiety Disorders; Depression; Behavior; Stereotyping; Cell Phone Use; Social Stigma

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of three intervention arms.
Who Masked: Participant, Outcomes Assessor
Masking Description: Random assignment to the 3 arms in a 1:1:1 allocation ratio will be determined centrally by the PI according to a random schedule. There is no practical way to blind the study participants to treatment and accomplish the objectives of the study. However, the study participants will be unaware of the aims of the arm to which they were assigned. Because they will not be blinded to the video exposure, the study participants assigned to one of the video contact arms will be aware that they are being exposed to a video-based contact intervention, and the study participants assigned to the waitlist control arm will be aware that they are being waitlisted. The research coordinator/team member (who will be conducting the outcome assessments) will be blinded to treatment assignment status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Video Intervention 1 (Experimental): The video intervention #1 will involve videos of patients describing personal narratives of mental illness, treatment and recovery, and will be delivered over 4 weeks (with two booster sessions in week 6 and 12). Assessments will be completed over 12 months from date of randomization.
  Interventions: Behavioral: Video Intervention 1
- Video Intervention 2 (Active Comparator): The video intervention #2 will involve videos of patients describing personal narratives of mental illness, treatment and recovery, and will be delivered over 4 weeks (with two booster sessions in week 6 and 12). Assessments will be completed over 12 months from date of randomization.
  Interventions: Behavioral: Video Intervention 2
- Waitlist Video Intervention 3 (Placebo Comparator): After the completion of the 6-month waitlist period, the experimental video intervention will be provided. The intervention will involve videos of patients describing personal narratives of mental illness, treatment and recovery, and will be delivered over 4 weeks (with two booster sessions in week 6 and 12). The intervention offered after the waitlist period will follow video intervention 1 (experimental arm).
  Interventions: Behavioral: Video Intervention 3

INTERVENTIONS:
Behavioral: Video Intervention 1 — A self-administered video-based mobile app with narratives on mental illness. The content of the videos consists of individuals sharing their personal experiences with depression and anxiety.
  Arms: Video Intervention 1
Behavioral: Video Intervention 2 — A self-administered video-based mobile app with narratives on mental illness. The content of the videos consists of individuals sharing their personal experiences with depression and anxiety.
  Arms: Video Intervention 2
Behavioral: Video Intervention 3 — An experimental self-administered video-based mobile app with narratives on mental illness after the waitlist period has been completed. The content of the videos consists of individuals sharing their personal experiences with depression and anxiety.
  Arms: Waitlist Video Intervention 3

SUMMARY:
Major depressive and anxiety disorders are highly prevalent in the general population and are a leading cause of disability. Black adults have a high burden of depression and anxiety. This study aims to assess a self- administered video-based intervention to reduce mental illness stigma and medical mistrust among Black adults with moderate to severe depression or anxiety.

DETAILED DESCRIPTION:
Major depressive and anxiety disorders affect 57.3 million adults in the U.S. These disorders are also highly stigmatized. Stigma refers to negative attitudes or beliefs about mental illness, or negative behaviors directed toward persons with mental illness (PWMI) is a leading and fundamental cause of health inequities.

The efficacy and precision of anti- stigma interventions to improve mental health outcomes among underserved Black adults are grossly limited and represent a critical public health gap. Studies show stigma compounds disabilities related to the primary symptoms of mental illness and increases morbidity and premature mortality related to mental illness. Compared with white adults, Black adults with mental illness have more chronic disease, and more severe illness at presentation. Meta-analyses have consistently shown that both face-to-face and video-based contact with individuals with mental illness can reduce stigma. Recent studies that distinguished contact delivery showed effect size for video-based contact to be comparable to face-to-face contact. Contact interventions, which are premised on the idea that positive and voluntary contact with PWMI can effectively reduce mental illness stigma, are aimed at reducing stigma and improving health outcomes.

The primary objective of this study is to evaluate the efficacy of a self-administered, video-based mobile app intervention aimed at reducing mental illness stigma among Black adults. Black adults with moderate to severe depression or anxiety will be recruited to participate in the Randomized Controlled Trial (RCT). Participants will be randomly assigned to one of three arms: two video-based intervention arms and one waitlist control arm. The video-based intervention will include first-hand lived experience stories of mental health and one's recovery journey.

ELIGIBILITY:
Inclusion Criteria:

1. If you identify as Black American or Black immigrant
2. Experience or been diagnosed with depression and/or anxiety
3. Age 18-45 years
4. Own a smartphone with internet access
5. Have not seen a psychiatrist or therapist in the last 12 months or have not been in routine healthcare
6. English speaking

Exclusion Criteria:

1. Visual, hearing, voice, or motor impairments that would prevent engagement in study procedures,
2. Diagnosis of psychotic disorder or severe suicidality for which participation would be inappropriate.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Treatment Inventory of Costs in Patients with Psychiatric Disorders | 12 months post intervention
  An adapted version to evaluate the utilization of mental health care services. The self-report questionnaire includes single item questions that will be used such as, "How many appointments have you attended at a Mental Health Care Institution in the past 3 months? Or at another mental health treatment facility?" and "In the past 3 months, how many appointments have you had with a psychologist, psychotherapist, or psychiatrist at a hospital?". Response options are qualitative: "no appointments" or providing the number of appointments attended. The test-retest reliability based on Cohen's Kappa was 0.649. Construct validity was assessed through the number of contacts recorded in the registration data, with a high correlation (ρ = 0.791).
Release of Information Form | 12 months post intervention
  The release of information form will be used to objectively measure the utilization of mental healthcare services by identifying visits made to these services. More or less visits is dependent on patient needs and does not have an intrinsic positive or negative value.

SECONDARY OUTCOMES:
Reported and Intended Behavior Scale | Pre-intervention and up to 12 months post-intervention
  The Reported and Intended Behavior Scale includes 4 questions on each of the reported and intended behaviors. Items 1-4 are binary, "yes" or "no". Items 5-8 are evaluated using a five-point Likert scale, ranging from 1 (strongly disagree) to 5 (strongly agree). The total score ranges from a minimum of 4 to a maximum of 20. Higher scores indicate less stigma (less desire for social distance) and lower scores indicate higher stigma (more desire for social distance). The test-retest reliability was 0.75, and internal consistency, based on Cronbach's alpha among items 5-8, was 0.85.
Internalized Stigma of Mental Illness | Pre-intervention and up to 12 months post-intervention
  The Internalized Stigma of Mental Illness is a 29-item measure with subscales that assess enacted and internalized stigma. Each item is evaluated using a four-point Likert scale, ranging from 1 (strongly disagree) to 4 (strongly agree). The total score ranges from a minimum of 29 to a maximum of 116. The higher scores indicate more internalized stigma. The original Internalized Stigma of Mental Illness reported test-retest reliability of 0.92.
The Group Based Medical Mistrust Scale | Pre-intervention and up to 12 months post-intervention
  The Group Based Medical Mistrust Scale is a 12 -item scale to measure race-based medical mistrust; it has strong validity and reliability. Each item is evaluated using a five-point Likert scale, ranging from 1 (strongly disagree) to 5 (strongly agree). The total score ranges from a minimum of 12 to a maximum of 60. Higher scores indicate greater medical mistrust.The Cronbach alpha for the full measure in previous studies was α=0.87-0.88. The total score and its three subscales were positively correlated with avoidance of health care (total score: p<0.0001; r=0.344).
Group Help Seeking Questionnaire | Pre-intervention and up to 12 months post-intervention
  The Group Help Seeking Questionnaire contains 10-items repeated for two problems (personal emotional and suicidal emotions). Each item is evaluated using a seven-point Likert scale, ranging from 1 (extremely unlikely) to 7 (extremely likely). The total score ranges from a minimum of 20 to a maximum of 140. Higher scores indicate higher help seeking intentions. Cronbach alpha for the full measure in previous studies was α=0.91. The perceived quality of previous mental health care was positively related to intentions to seek help from a mental health professional for personal-emotional problems, rs(55) = 0.51, p < 0.001, and suicidal thoughts, rs(54) = 0.57, p < 0.001.

CONTACTS AND LOCATIONS:
Overall Officials: Aderonke Pederson, MD, Principal Investigator — Massachuessets General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bouwmans C, De Jong K, Timman R, Zijlstra-Vlasveld M, Van der Feltz-Cornelis C, Tan Swan S, Hakkaart-van Roijen L. Feasibility, reliability and validity of a questionnaire on healthcare consumption and productivity loss in patients with a psychiatric disorder (TiC-P). BMC Health Serv Res. 2013 Jun 15;13:217. doi: 10.1186/1472-6963-13-217. PMID 23768141
- [Background] Boyd JE, Adler EP, Otilingam PG, Peters T. Internalized Stigma of Mental Illness (ISMI) scale: a multinational review. Compr Psychiatry. 2014 Jan;55(1):221-31. doi: 10.1016/j.comppsych.2013.06.005. Epub 2013 Sep 21. PMID 24060237
- [Background] Evans-Lacko S, Rose D, Little K, Flach C, Rhydderch D, Henderson C, Thornicroft G. Development and psychometric properties of the reported and intended behaviour scale (RIBS): a stigma-related behaviour measure. Epidemiol Psychiatr Sci. 2011 Sep;20(3):263-71. doi: 10.1017/s2045796011000308. PMID 21922969
- [Background] Ibrahim N, Amit N, Shahar S, Wee LH, Ismail R, Khairuddin R, Siau CS, Safien AM. Do depression literacy, mental illness beliefs and stigma influence mental health help-seeking attitude? A cross-sectional study of secondary school and university students from B40 households in Malaysia. BMC Public Health. 2019 Jun 13;19(Suppl 4):544. doi: 10.1186/s12889-019-6862-6. PMID 31196033
- [Background] Thompson HS, Valdimarsdottir HB, Winkel G, Jandorf L, Redd W. The Group-Based Medical Mistrust Scale: psychometric properties and association with breast cancer screening. Prev Med. 2004 Feb;38(2):209-18. doi: 10.1016/j.ypmed.2003.09.041. PMID 14715214